CLINICAL TRIAL: NCT02349269
Title: Postoperative Atrial Fibrillation After Cardiac Surgery is Not an Independent Risk Factor for Long-term Cardiovascular Morbidity and Mortality in Anticoagulated Patients
Brief Title: Postoperative Atrial Fibrillation and Long-term Survival
Acronym: POAF
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Other Study IDs: samuelm1
Record Dates: First submitted 2014-12-01; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2014-11

CONDITIONS: Death; Stroke; Myocardial Infarction
Keywords: Atrial fibrillation; CABG; Stroke
MeSH Terms: conditions — Death; Stroke; Myocardial Infarction; Atrial Fibrillation

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 105 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the investigators trial was to evaluate association between new onset postoperative atrial fibrillation (POAF) and late cardiovascular morbidity and mortality.

DETAILED DESCRIPTION:
The material of this retrospective study consist patients without preoperative history of atrial fibrillation, participated in three different randomized controlled trials previously . A total of 519 consecutive patients underwent coronary artery bypass surgery, aortic valve replacement or combined aortic valve with coronary bypass surgery in Kuopio University Hospital from 2004 to 2008. Patients with previous episodes of atrial fibrillation (AF) or flutter and also patients with mitral valve surgery were excluded. All patients had continuous postoperative ECG monitoring for at least 48 hours. AF episodes lasting longer than 5 minutes were registered. Thereafter 12 lead ECG was recorded daily and in case of symptoms of rhythm disturbances.

Medical records were reviewed during 2012 using standardized data collection protocol. Statistics Finland database was used for mortality data.

ELIGIBILITY:
Inclusion Criteria:

* previously cardiac operation, CABG or AVR

Exclusion Criteria:

* Previous Atrial fibrillation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients without preoperative history of atrial fibrillation, participated in three different randomized controlled trials previously
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
cardiovascular and all-cause death | 1-105 month
stroke | 1-105 month
late atrial fibrillation | 1-105 month
myocardial infarction | 1-105 month